CLINICAL TRIAL: NCT03112876
Title: Sebum Collection for Analysis and Correlation to Sebum Production, Barrier Function, and With Cutaneous and Internal Inflammatory Disease
Brief Title: Sebum Collection and Skin Barrier Function Analysis
Acronym: Sebum
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 605131
Record Dates: First submitted 2014-07-10; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Smoking; Acne; Atopic Dermatitis; Aging
Keywords: younger age; older age; atopic dermatitis; acne; smoker
MeSH Terms: conditions — Smoking; Acne Vulgaris; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Young Age - Healthy: These subjects are between the age of 12 and 35 years. This group will undergo the following intervention: skin surface lipid collection via tapes and skin barrier function evaluated with non-invasive painless devices.
  Interventions: Other: Skin Surface Lipid Collection and Skin Barrier Function
- Old Age -Healthy: These subjects are 55 years of age and older. This group will undergo the following intervention: skin surface lipid collection via tapes and skin barrier function evaluated with non-invasive painless devices.
  Interventions: Other: Skin Surface Lipid Collection and Skin Barrier Function
- Active Smoker: These subjects are active smokers who smoke often. This group will undergo the following intervention: skin surface lipid collection via tapes and skin barrier function evaluated with non-invasive painless devices.
  Interventions: Other: Skin Surface Lipid Collection and Skin Barrier Function
- Dermatological skin condition: Acne vulgaris: These subjects have acne vulgaris. This group will undergo the following intervention: skin surface lipid collection via tapes and skin barrier function evaluated with non-invasive painless devices.
  Interventions: Other: Skin Surface Lipid Collection and Skin Barrier Function
- Dermatological skin condition: Atopic dermatitis: These subjects have atopic dermatitis. This group will undergo the following intervention: skin surface lipid collection via tapes and skin barrier function evaluated with non-invasive painless devices.
  Interventions: Other: Skin Surface Lipid Collection and Skin Barrier Function

INTERVENTIONS:
Other: Skin Surface Lipid Collection and Skin Barrier Function — All five groups will undergo the same study intervention: skin surface lipid collection via tapes and skin barrier function evaluated with non-invasive painless devices.
  Other Names: lipid profile; sebum secretion rate; skin water loss; skin hydration

SUMMARY:
The goal is this study is to evaluate how the skin surface lipid composition is correlated with overall sebum production, barrier function, and inflammatory disease status. We hypothesize that there will be differences in the skin surface composition among subjects of various groups:

1. Young vs older healthy population
2. Atopic dermatitis vs Acne vs Healthy controls
3. Active smokers vs non-smoker controls

DETAILED DESCRIPTION:
This study will be conducted through the use of painless tapes to collect lipid. These will be applied to the skin and removed. Secondly, the barrier function will be evaluated through the use of non-invasive painless devices that measure sebum, skin water loss, and skin hydration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that are 12 years of age or older

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study patients will be recruited from the UC Davis Department of Dermatology, UC Davis undergraduate campus, Sacramento State University, and from the greater Sacramento area.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2016-02-26 (Actual); Study Completion 2016-02-26 (Actual)

PRIMARY OUTCOMES:
Lipid Profile-aging | 1 day
  The lipid profile of the subject group will be evaluated through the use of painless tapes that will be applied to the skin.
Lipid Profile-acne | 1 day
  The lipid profile of the subject group will be evaluated through the use of painless tapes that will be applied to the skin.
Lipid Profile-atopic dermatitis | 1 day
  The lipid profile of the subject group will be evaluated through the use of painless tapes that will be applied to the skin.
Lipid Profile-smoking | 1 day
  The lipid profile of the subject group will be evaluated through the use of painless tapes that will be applied to the skin.

SECONDARY OUTCOMES:
Skin Barrier Function- aging | 1 day
  The skin barrier function will be evaluated for this group through the use of non-invasive handheld devices. These devices provide information about sebum secretion rate, skin water loss, and skin hydration.
Skin Barrier Function- acne | 1 day
  The skin barrier function will be evaluated for this group through the use of non-invasive handheld devices. These devices provide information about sebum secretion rate, skin water loss, and skin hydration.
Skin Barrier Function- atopic dermatitis | 1 day
  The skin barrier function will be evaluated for this group through the use of non-invasive handheld devices. These devices provide information about sebum secretion rate, skin water loss, and skin hydration.
Skin Barrier Function- smoking | 1 day
  The skin barrier function will be evaluated for this group through the use of non-invasive handheld devices. These devices provide information about sebum secretion rate, skin water loss, and skin hydration.

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Department of Dermatology, Sacramento, California, United States

REFERENCES:
- [Background] Ni Raghallaigh S, Bender K, Lacey N, Brennan L, Powell FC. The fatty acid profile of the skin surface lipid layer in papulopustular rosacea. Br J Dermatol. 2012 Feb;166(2):279-87. doi: 10.1111/j.1365-2133.2011.10662.x. PMID 21967555
- [Background] Sakai S, Kikuchi K, Satoh J, Tagami H, Inoue S. Functional properties of the stratum corneum in patients with diabetes mellitus: similarities to senile xerosis. Br J Dermatol. 2005 Aug;153(2):319-23. doi: 10.1111/j.1365-2133.2005.06756.x. PMID 16086742
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical